CLINICAL TRIAL: NCT01876862
Title: A Pilot Study Evaluating the Maintenance of Viral Suppression After 24 Weeks of Therapeutic Interruption in Chronically HIV-1 Infected Patients With a Low Circulating HIV-DNA Reservoir
Brief Title: Towards HIV Functional Cure
Acronym: ULTRASTOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Objectif Recherche Vaccins SIDA (Other)
Collaborators: Fondation Bettencourt-Schueller (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ORVACS 012
Record Dates: First submitted 2013-05-31; First posted 2013-06-13 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Chronic HIV-1 Infection
Keywords: HIV-1; chronic infection; cure; remission
MeSH Terms: conditions — Persistent Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- STOP ART (Experimental): Antiretroviral treatment interruption in 3 successive groups of 5 patients.
  "Zero-risk" strategy If after 8 weeks of treatment interruption, at least 1 patient from group 1 does not present any of the failure criteria, patients from group 2 will be included and their treatment interrupted. If after 8 weeks of treatment interruption, at least 2 patients from groups 1 and 2 do not present any failure criteria, patients from group 3 will be included and their treatment interrupted.
  Interventions: Other: Antiretroviral treatment interruption

INTERVENTIONS:
Other: Antiretroviral treatment interruption — pilot study in chronically HIV-infected patients with an ultralow HIV reservoir undergoing treatment-interruption.

SUMMARY:
During the ERAMUNE-01 and -02 studies, the HIV-DNA quantification in the PBMCs (Peripheral Blood Mononuclear Cells) showed showed that some patients had a very low or undetectable reservoir.

Recent studies showed that a low reservoir is associated to a spontaneous virologic control in three specific categories of patients:

* "Elite Controllers": these rare patients are able to spontaneously maintain an HIV-RNA viral load below 50 copies/mL and elevated CD4 counts without any treatment. These patients belong to the B27/B57 haplotypes associated to a reduced risk of HIV contamination but these haplotypes are very rare in the global population (0,3 %)
* "Visconti" patients: early-treated patients, during the primo-infection stage. After 3 to 5 years of treatment, these patients are able to maintain an undetectable HIV-RNA viral load.
* "Salto" patients: these patients are treated a bit later compared to the Visconti cohort, when their CD4 count was above 350 cells/mm3 and their HIV-RNA viral load below 50 000 copies/mL. The follow-up of these patients showed the same capacity of control of the HIV infection for at least 2 years following treatment interruption.

Taking into account these 3 categories of patients which common characteristics is a low reservoir, our objective is to answer the 2 following questions:

1. Is it possible to discontinue the treatment in chronically-infected patients with a "normal" immune system and with an undetectable HIV-DNA reservoir?
2. Is a low viral reservoir predictive of a treatment-free remission of the HIV infection in chronically-infected patients?

The main objective of the proof-of-concept ERAMUNE-03 trial is to evaluate the proportion of patients in success (i.e. able to maintain a virologic and an immunologic control of the infection) after treatment discontinuation, failure is defined as:

* An HIV-RNA viral load > 400 copies/mL on 2 consecutive tests starting from Week 4
* Or CD4 count < 400 cells/mm3 on 2 consecutive measures starting from Week 4
* Or the onset of an AIDS-related event

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected patient
* CD4 count > 500 cells/mm3
* CD4/CD8 ratio > 0.9
* CD4 nadir > 300 cells/mm3
* HIV-1-RNA plasma viral load < 50 copies/mL under antiretroviral treatment for at least 2 years
* HIV-1-RNA plasma viral load < 20 copies/mL at baseline
* HIV-DNA reservoir < 100 copies/million PBMCs
* Signed fully informed consent form
* Ability to attend the complete schedule of assessments and patient visits
* Patient eligible for national social insurance

Exclusion Criteria:

* Medical history of AIDS-staging event
* Antiretroviral treatment initiated during primo-infection in absence of anti-HIV antibodies (negative ELISA and Western Blot tests)
* Change in the antiretroviral treatment combination within the 3 months prior inclusion
* HIV-2 co-infection
* History of thrombocytopenia (< 100 000 cells/mm3)
* Acute neurologic event during primo-infection
* Chronic and active hepatitis B as defined as positive HBs antigen or positive isolated anti-HBc antibodies
* Chronic and active hepatitis C as defined as positive anti-HCV antibodies and positive HCV-RNA PCR
* History of cancer within the 5 years prior inclusion except basocellular cutaneous cancers
* Comorbidity associated to lifespan < 12 months according investigator's opinion
* History of auto-immune disease (lupus erythematous, Hashimoto's thyroiditis, ...)
* Hemoglobin < 7 g/dL, Creatinine clearance < 60 mL/min using the MDRD formula
* Patients refusal to use a condom for any sexual relationship during the course of the study
* Refusal from women of childbearing potential to use at least one additional barrier method other than condoms
* Ongoing pregnancy as documented by a positive blood test performed at screening or later
* Lactating woman
* Psychologic unstability or patient state-of-mind incompatible with the participation in the study as evaluated by psychologist at screening
* Drug or alcohol addiction or abuse
* Concomitant participation to another trial involving any investigational treatment or device

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in success | Week 24
  Success is defined as the maintenance of the controlled viral infection after 24 weeks of therapeutic interruption. Failure is defined as:
  * An HIV-1-RNA plasma viral load > 400 copies/mL starting from Week 4 as confirmed by two consecutive measures within 2 to 4 weeks
  * Or a CD4 count < 400 cells/mm3 starting from Week 4 as confirmed by two consecutive measure within 2 to 4 weeks
  * Or the onset of an AIDS-grading clinical event (grade B or C in the CDC classification, version 1993)

SECONDARY OUTCOMES:
Changes from baseline in CD4 and CD8 lymphocytes counts | Up to Week 48
Changes from baseline in immune activation and inflammation markers | Up to Week 48
Changes from baseline in anti-HIV specific T cells response | Up to Week 48
Quantitative and qualitative changes from baseline in the HIV-1 reservoir as measured on sorted CD4 lymphocytes subsets | Up to Week 48
  CD4 subpopulations will be live-sorted and purified. In each subset defined by surface markers, HIV-1 DNA will be quantified and transcriptional potential of HIV will be evaluated.
Proportion of patients in virologic success (HIV-1-RNA plasma viral load < 400 copies/mL) | Up to Week 48
Changes from baseline in the HIV-1 reservoir as measured by HIV-1 DNA copies per million PBMCs | Up to Week 48
Changes from baseline in the proportion of defective HIV-1 DNA | Up to Week 48
  Evaluation of the stop codons in the HIV-1 DNA sequence
Changes from baseline in the plasma concentrations of antiretroviral molecules | Up to Week 48
Changes from baseline in the patient quality of life and in the disease-related symptoms | Up to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: François LECARDONNEL, MSc, Study Director — Objectif Recherche Vaccins SIDA; Christine KATLAMA, MD, Principal Investigator — Hospital Pitié-Salpêtrière
Locations (2):
- France (2):
  - University Hospital of Bicêtre, Le Kremlin-Bicêtre
  - Hospital Pitié-Salpêtrière, Paris